CLINICAL TRIAL: NCT01163942
Title: A RANDOMIZED CONTROLLED STUDY IN NEWLY DIAGNOSED SEVERE APLASTIC ANEMIA PATIENTS RECEIVING ANTITHYMOCYTE GLOBULIN (ATG), CYCLOSPORIN A, WITH OR WITHOUT G-CSF
Brief Title: Randomized Study In Severe Aplastic Anemia Patients Receiving Atg, Cyclosporin A, With Or Without G-CSF (SAA-G-CSF)
Acronym: SAA-G-CSF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Ceased production of the study drug, Lymphoglobulin. Recruitment of patients onto the trial was too slow.
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Flagship AA trial; 41980964 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Aplastic Anaemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No G-CSF, No 2nd ATG (Active Comparator): Patients randomised not to receive G-CSF (alongside ATG and CSA) and to not receive early retreatment in case of no response.
  Interventions: Drug: G-CSF; Drug: Early retreatment with ATG
- No G-CSF, yes 2nd ATG (Active Comparator): Patients randomised not to receive G-CSF (alongside ATG and CSA) but they do receive early retreatment in case of no response.
  Interventions: Drug: G-CSF; Drug: Early retreatment with ATG
- Yes G-CSF, No 2nd ATG (Active Comparator): Patients randomised to receive G-CSF (alongside ATG and CSA) and to not receive early retreatment in case of no response.
  Interventions: Drug: G-CSF; Drug: Early retreatment with ATG
- Yes G-CSF, Yes 2nd ATG (Active Comparator): Patients randomised to receive G-CSF (alongside ATG and CSA) and to receive early retreatment in case of no response.
  Interventions: Drug: G-CSF; Drug: Early retreatment with ATG

INTERVENTIONS:
Drug: G-CSF — Yes/no addition of G-CSF
Drug: Early retreatment with ATG — Yes/no early retreatment with ATG

SUMMARY:
The purpose of this study is to examine the effect of G-CSF on disease free survival and overall survival in aplastic anaemia patients who also receive ATG and Cyclosporin A.

DETAILED DESCRIPTION:
Open label, randomized, controlled study of G-CSF, ATG and Cyclosporin A versus ATG and Cyclosporin A. Subjects will be evaluated for hematologic response through day 240. Subjects who do not demonstrate a partial or complete remission by day 120 will be randomized to receive either a second course of ATG or continue their current regimen. Subjects who do demonstrate a partial or complete remission will continue their current regimen through day 240 or maintenance of a complete remission for 30 days. The last day of study treatment will be day 240.

ELIGIBILITY:
Inclusion Criteria:

* Severe or very severe aplastic anemia
* Less than 6 months from diagnosis of severe aplastic anemia by bone marrow biopsy
* Ethical - Before randomization is done the subject or legally acceptable representative must give written informed consent for participation in the study

Exclusion Criteria:

* Eligibility for an HLA-matched sibling donor transplant
* Prior therapy with ATG
* Cyclosporin A <4 weeks before enrollment
* Treatment with G-CSF <2 weeks before enrollment
* Other growth factors <4 weeks before enrollment
* Diagnosis of Fanconi anemia, dyskeratosis congenita or congenital bone marrow failure syndrome
* Evidence of myelodysplastic disease
* Diagnosis or previous history of carcinoma (except local cervical, basal cell, squamous cells, or melanoma)
* Subjects who have infection, hepatic, renal cardiac, metabolic or other concurrent diseases of such severity that death is imminent
* Subject is pregnant (e.g. positive HCG test) or is breast feeding

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2001-03; Primary Completion 2008-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Failure free survival | day 240
  To evaluate the effect of G-CSF on failure free survival and mortality in study subjects also receiving ATG and Cyclosporin A & time to hematologic response (failure defined as death, non-response or requirement of further treatment).

SECONDARY OUTCOMES:
Haematological response | day 240
  The proportion of subjects who achieve a hematologic response
Severe Infections | day 240
  Incidence of severe infections
Benefit of addition of G-CSF | day 240
  The benefit due to the addition of G-CSF on death rate (i), days of hospitalization (ii), and duration of antibiotic treatment (iii)
Complete remission | day 120
  Time to achieving a complete remission within 120 days
Relapse rate | 2year
  The relapse rate among responders
Blood count | day 240
  Median blood counts among subjects who achieve transfusion independence
Severity of the disease | day 365
  The proportion of subjects who have a change in severity of disease (e.g. improvement from very severe to severe aplastic anemia)
Retreatment with ATG | day 240
  Proportion of subjects who respond to re-treatment with ATG,
Safety | 6year
  The safety of G-CSF in subjects treated with G-CSF, ATG and Cyclosporin A, compared to subjects who receive ATG and Cyclosporin A

CONTACTS AND LOCATIONS:
Overall Officials: André Tichelli, Prof. MD., Principal Investigator — University Hospital, Basel, Switzerland
Locations (71):
- University Hospital, Pilsen, Czechia
- France (16):
  - CHU Angers, Angers
  - Avicenne Hospital, Bobigny
  - University Hospital, Brest
  - CHU Clemenceau, Caen
  - CHU de Caen, Caen
  - Henri Mondor, Créteil
  - CHU Limoges, Limoges
  - Paoli-Calmettes Institute, Marseille
  - CHU Montpellier, Montpellier
  - CHU Caremeau, Nîmes
  - St. Antoine, Paris
  - St. Louis Hospital, Paris
  - CHU Reims, Reims
  - CHU Toulouse, Toulouse
  - Bretonneau Hospital, Tours
  - G. Roussy Institute, Villejuf
- Germany (33):
  - Benjamin Franklin Hospital, Berlin
  - Charite Hospital, Berlin
  - Evangelisches Waldkrankenhaus, Berlin
  - Evangelisches Krankenhaus Diakonie, Bremen
  - University Hospital, Cologne
  - University Hospital Carl Gustav Carus, Dresden
  - St. Johannes-Hospital, Duisburg
  - University Hospital Heinrich Heine, Düsseldorf
  - Universitätsklinik, Essen
  - University Hospital, Frankfurt
  - University Hospital Georg August, Göttingen
  - Marien Hopistal, Hagen
  - University Hospital, Halle
  - Asklepios Klinik Altona, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital, Heidelberg
  - Universitäts Klinikum, Ludwigshaven
  - Sana Klinikum, Lübeck
  - Harlachin, München
  - Klinkum Rechts der Isar, München
  - Krakenhaus München Schwabing, München
  - Klinikum Nord, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Brüderkrankenhaus St. Josef, Paderborn
  - Klinikum Ernst von Bergmann, Potsdam
  - University Hospital, Regensburg
  - University Hospital, Rostock
  - Klinikum Stuttgart, Stuttgart
  - University Clinic Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - Deutsche Klinik für Diagnostik, Wiesbaden
  - University Hospital, Wiesbaden
  - Helios Klinikum Wuppertal, Wuppertal
- Greece (2):
  - Athens General Pediatric Hospital, Athens
  - University Hospital, Pátrai
- Italy (4):
  - Gaslini Children's Hospital, Genova
  - San Martino, Genova
  - San Raffaele Hospital, Milan
  - University Hospital, Padua
- Netherlands (3):
  - Groningen University Hospital, Groningen
  - Leiden University Medical Centre, Leiden
  - Erasmus MC, Rotterdam
- Sweden (2):
  - Lund Unversity, Lund
  - Huddinge University Hospital, Stockholm
- Switzerland (2):
  - University Hospital, Basel
  - Hopitaux Universitaires de Geneve, Geneva
- United Kingdom (8):
  - Monklands Hospital, Airdrie
  - Heartlands Hospital, Birmingham
  - Bristol Haematology & Oncology Centre, Bristol
  - Royal Cornwall Hospitals, Cornwall
  - The Leeds Teaching Hospitals, Leeds
  - St George's Hospital/ St George's University of London, London
  - St. Bartholomew's Hospital, London
  - Wishaw General, Wishaw

REFERENCES:
- [Derived] Tichelli A, de Latour RP, Passweg J, Knol-Bout C, Socie G, Marsh J, Schrezenmeier H, Hochsmann B, Bacigalupo A, Samarasinghe S, Rovo A, Kulasekararaj A, Roth A, Eikema DJ, Bosman P, Bader P, Risitano A, Dufour C; SAA Working Party of the EBMT. Long-term outcome of a randomized controlled study in patients with newly diagnosed severe aplastic anemia treated with antithymocyte globulin and cyclosporine, with or without granulocyte colony-stimulating factor: a Severe Aplastic Anemia Working Party Trial from the European Group of Blood and Marrow Transplantation. Haematologica. 2020 May;105(5):1223-1231. doi: 10.3324/haematol.2019.222562. Epub 2019 Oct 3. PMID 31582549
- [Derived] Tichelli A, Schrezenmeier H, Socie G, Marsh J, Bacigalupo A, Duhrsen U, Franzke A, Hallek M, Thiel E, Wilhelm M, Hochsmann B, Barrois A, Champion K, Passweg JR. A randomized controlled study in patients with newly diagnosed severe aplastic anemia receiving antithymocyte globulin (ATG), cyclosporine, with or without G-CSF: a study of the SAA Working Party of the European Group for Blood and Marrow Transplantation. Blood. 2011 Apr 28;117(17):4434-41. doi: 10.1182/blood-2010-08-304071. Epub 2011 Jan 13. PMID 21233311